CLINICAL TRIAL: NCT03189628
Title: Study of Autologous Stromal Vascular Fraction From Adipose Tissue in Promoting Skin Regeneration
Brief Title: The Effect of Autologous Stromal Vascular Fractions on Skin Regeneration
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, MD, PhD, Professor, Head of Departement of Plastic and Reconstructive Surgery, Shanghai 9th People's Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-261-T196
Record Dates: First submitted 2017-05-22; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Skin; Aging
Keywords: stromal vascular fraction; skin regeneration; skin texture; anti-aging
MeSH Terms: interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stromal vascular fraction (Experimental): Transplantation of resuspended SVF
  Interventions: Biological: stromal vascular fraction
- saline (Placebo Comparator): 1 ml saline without cells will be used as placebo.
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: stromal vascular fraction — The adipose tissue(no less than 40ml) in abdomen will be harvested and digested at 37 °C for (45-60) min with (0.125-1.5)mg/ml collagenase . After filtration and centrifugation at the speed of (700-1500)g, mature adipocytes are separated from the cell pellet. The pellet then is treated with saline twice to remove cell fragment and rudimental collagenase . The harvested pellet is stromal vascular fraction (SVF) The SVF was resuspended in 1 ml saline and transplanted for 3 area including the forehead、palpebra inferior and crow's-feet.
  Other Names: heterogeneous cell populations isolated from adipose tissue
  Arms: stromal vascular fraction
Drug: Saline — 1 ml saline was injected for 3 area including the forehead、palpebra inferior and crow's-feet.
  Other Names: normal saline
  Arms: saline

SUMMARY:
The purpose of this study is to observe whether the transplantation of autologous stromal vascular fraction (SVF) in adipose tissue is safe and its effect on improving skin regeneration.

DETAILED DESCRIPTION:
This is a randomized controlled single blind clinal trial that designed to observe whether the transplantation of autologous stromal vascular fraction (SVF) in adipose tissue is safe and its effect on improving skin regeneration.

The clinical trial will concentrate on the therapeutic effect of SVF after facial injection. After 1, 4, 8, 12, 24 and 48 weeks of treatment, a comprehensive examination of the facial skin was performed to assess the effect of the SVF. Skin texture, thickness and colour will be observed to evaluate the effect of SVF on skin regeneration

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 65.
* No other facial plastic surgery or cosmetic surgery was performed during the study period (frontal, temporal, and lower eyelid).
* Intends to undergo facial anti-aging treatment with SVF

Exclusion Criteria:

* Not fit for stem cells graft treatment.
* Evidence of infection, ischemia, ulcer or other pathological changes within the targeting area which defined as not suitable for SVF treatment; or history of delayed healing, radiational therapy.
* Significant renal, cardiovascular, hepatic and psychiatric diseases.
* Significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV).
* Used external medication on the targeting area within 4 weeks.
* Skin invasive treatment including laser on the targeting area within 6 months.
* Hyaluronic acid injection on the targeting area within 12 months.
* Botulinum toxin injection on the targeting area within 6 months.
* History of any hematological disease, including leukopenia , thrombocytopenia, or thrombocytosis.
* Evidence of malignant diseases or unwillingness to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-08-25 (Estimated); Study Completion 2018-03-13 (Estimated)

PRIMARY OUTCOMES:
Measure the texture changes of the skin | Baseline and 12 months post the treatment
  Using Cutometer® dual MPA 580 in 12 months post the treatment.

SECONDARY OUTCOMES:
Measure the colour changes of the skin | Baseline and 12 months post the treatment
  Using Canfield Scientific VISIA in 12 months post the treatment.
Occurence of major adverse events | Up to approximately 12 months after study start
  Including skin necrosis, infection, erythra and all other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Li Qingfeng, MD; PhD, Study Chair — Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Qin J, Cheng C, Huang RL, He J, Zhou S, Tan PC, Zhang T, Fang B, Li Q, Xie Y. Isolation of the Stromal Vascular Fraction Using a New Protocol with All Clinical-Grade Drugs: From Basic Study to Clinical Application. Aesthetic Plast Surg. 2024 Nov;48(22):4702-4711. doi: 10.1007/s00266-024-04221-9. Epub 2024 Jul 10. PMID 38987318